CLINICAL TRIAL: NCT03892499
Title: An Open-label, 2-Period, Fixed-sequence, Phase 1 Study in Healthy Volunteers to Evaluate the Effect of Itraconazole, a Potent CYP3A Inhibitor, on the Pharmacokinetics of Olinciguat (IW-1701)
Brief Title: A Trial to Evaluate the Effect of Itraconazole (ITZ), a CYP3A4 Inhibitor, on the Pharmacokinetics of the Soluble Guanylate Cyclase Stimulator, Olinciguat (IW-1701), in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cyclerion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OLI-105
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental): Period 1: Single dose of olinciguat. Period 2: ITZ is dosed once daily (QD) for 10 days; a single dose of olinciguat is administered 1 hour after the fourth ITZ QD dose.
  Interventions: Drug: Olinciguat; Drug: Itraconazole

INTERVENTIONS:
Drug: Olinciguat — Oral Tablet
  Other Names: IW-1701
Drug: Itraconazole — Oral Capsule

SUMMARY:
To evaluate the effect of itraconazole (a potent cytochrome P450 isoenzyme [CYP]3A inhibitor) on the pharmacokinetics (PK) of olinciguat

ELIGIBILITY:
Inclusion Criteria:

* Subject is an ambulatory adult and between 18 and 55 years old (inclusive) at the screening visit
* Subject is in good health and has no clinically significant findings on physical examination
* Body mass index is > 18 and < 30 kg/m2 at the screening visit
* Women of reproductive potential must have a negative pregnancy test at screening at at the time of check-in and must agree to use protocol-specified contraception throughout the duration of the study and until 90 days after receiving the final study drug dose
* Men must agree to use protocol-specified contraception and also to not donate sperm throughout the study and until 90 days after receiving the final study drug dose
* Other inclusion criteria per protocol

Exclusion Criteria:

* Any active or unstable clinically significant medical condition
* Use of any prescribed or non-prescribed medication (except for hormonal birth control)
* Other exclusion criteria per protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2019-06-23 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of olinciguat | Predose and up to 8 days post first olinciguat dose
Area under the plasma concentration time curve from time zero (predose) extrapolated to infinity (AUCinf) | Predose and up to 8 days post first olinciguat dose

SECONDARY OUTCOMES:
Number of subjects with ≥1 treatment-emergent adverse event (TEAE) in Period 1 vs Period 2 | 51 days post first olinciguat dose
Cmax of Itraconazole | First Itraconazole dose up to day 8 of Period 2 (Period 2 duration can be up to 13 days)
Area under the concentration-time curve during a dosing interval (AUCtau) for itraconazole and hydroxy-itraconazole | Period 2 (Period 2 duration can be up to 13 days) predose and up to 24 hour after 2nd olinciguat dose
Cmax of hydroxy-Itraconazole | First Itraconazole dose up to day 8 of Period 2 (Period 2 duration can be up to 13 days)

CONTACTS AND LOCATIONS:
Overall Officials: Bina Tejura, MD, Study Director — Cyclerion Therapeutics
Locations (1):
- PPD, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No